CLINICAL TRIAL: NCT05094492
Title: Evaluation of Remineralization Potential of Self Assembling Peptide P11-4 Combined With Fluoride Compared to Fluoride Varnish in Management of Incipient Carious Lesions Using Laser Fluorescence: Randomized Clinical Trial
Brief Title: Evaluation of Remineralization Potential of Self Assembling Peptide Combined With Fluoride
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p11-4
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Caries; Initial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self assembling peptide P11-4 with fluoride (Experimental): P11-4 forms a 3D matrix within subsurface of incipient carious lesions , allowing formation of new hydroxyapatite crystal facilitating guided regeneration of enamel lesions. Combination with fluoride will have a synergistic effect on remineralization potential
  Interventions: Combination Product: Curodont Repair Fluoride Plus
- Fluoride varnish (Active Comparator): Gold standard agent for remineralization of incipient carious lesions.
  Interventions: Other: Bifluorid 10 fluoride varnish

INTERVENTIONS:
Combination Product: Curodont Repair Fluoride Plus — P11-4 self assembling peptide combined with fluoride
  Arms: Self assembling peptide P11-4 with fluoride
Other: Bifluorid 10 fluoride varnish — 5% Sodium Fluoride varnish (equal to 22,600 ppm fluoride)
  Arms: Fluoride varnish

SUMMARY:
Self-assembling peptide (P11-4) exhibited an outstanding ability for biomimetic re-mineralization of incipient enamel carious lesions. It creates a 3D matrix within the subsurface of carious lesions, allowing de novo formation of Hydroxyapatite crystals, thus enabling guided enamel regeneration of the demineralized enamel structure. Addition of fluoride to P11-4 may have a synergistic effect on the remineralization potential.

DETAILED DESCRIPTION:
This study is a randomized clinical trial, with parallel study design, 1:1 allocation ratio and superiority framework. The aim of the current trial is to evaluate remineralization potential of P11-4 combined with fluoride compared to fluoride varnish in management of incipient white spot carious lesions. Progress of the lesions will be assessed using laser fluorescence (DIAGNOdent).

ELIGIBILITY:
Inclusion Criteria:

* Active carious white spot lesions.
* Patient compliance.
* Controlled oral hygiene condition.

Exclusion Criteria:

* Participant in another trial.
* Non carious lesions.
* Systemic diseases or concomitant medication affecting salivary flow.
* Cavitation of carious lesions.
* Parafunctional habits.
* Pregnancy.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Remineralization | 6 months
  measuring carious lesion development using DIAGNOdent laser fluorescence (scores from 0 to 99) according to progression of the carious lesion

CONTACTS AND LOCATIONS:
Overall Officials: Omar O Shaalan, PhD, Principal Investigator — Lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No